CLINICAL TRIAL: NCT02936479
Title: Use of C1-INH (Berinert) for Renal Allograft Salvage in Refractory Antibody Mediated Rejection
Brief Title: C1-Inhibitor (INH) for Refractory Antibody Mediated Renal Allograft Rejection
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: CSL Behring (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 16-01851
Record Dates: First submitted 2016-10-14; First posted 2016-10-18 (Estimated); Results first posted 2019-07-11 (Actual); Last update posted 2019-07-11 (Actual); Status verified 2019-07

CONDITIONS: Antibody Mediated Rejection of Kidney Transplant
MeSH Terms: interventions — Complement C1 Inhibitor Protein

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Berinert treatment (Experimental)
  Interventions: Drug: C1-INH (Berinert)

INTERVENTIONS:
Drug: C1-INH (Berinert)

SUMMARY:
This is an open-label, single arm trial in which patient who have ongoing antibody mediated rejection of a kidney transplant deemed refractory to maximal medical therapy are given the complement inhibitor C1-INH (Berinert) in an effort to protect the graft from ongoing antibody mediated injury. A maximum of 5 patients will be enrolled.

ELIGIBILITY:
Inclusion Criteria:

* Kidney transplant with acute antibody mediated rejection refractory to standard therapy

Exclusion Criteria:

* Patients with known intolerance of or anaphylaxis to Berinert

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2018-10-30 (Actual); Study Completion 2018-10-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Montgomery, MD, Principal Investigator — NYU Langone Health
Locations (1):
- New York University School of Medicine, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Berinert Treatment: C1-Inhibitor (INH) (Berinert): C1 esterase inhibitor, Berinert, 25-50 units/kg, intravenous, 7 doses on days 1, 3, 5, 7, 9, 11, 13 and 50 units/kg twice weekly for a total study period of 6 months.
Period: Overall Study
Arm/Group | Berinert Treatment
Started | 1
Completed | 1
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Berinert Treatment: C1-INH (Berinert)
Arm/Group | Berinert Treatment
Number analyzed (Participants) | 1
Age, Customized [Count of Participants; unit: Participants]
  54 Years Old | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 1
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 1

OUTCOME MEASURES:

1. Primary Outcome: Renal Allograft Survival Measured by Severe and Refractory Antibody Mediated Renal (AMR)
Description: number of patients that presented with severe and refractory Antibody Mediated Renal (AMR) following kidney transplant and survived beyond one year after study drug administration
Time Frame: 24 months
Measure: Count of Participants; unit: Participants
Arm/Group | Berinert Treatment
Number analyzed (Participants) | 1
Participants | 1

ADVERSE EVENTS:
Time Frame: 17 months
Arm/Group | Berinert Treatment
All-Cause Mortality (participants affected / at risk) | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 1/1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Berinert Treatment (N=1)
skin infection (Skin and subcutaneous tissue disorders) | 1 (1) — left posterior extremity skin infection
urinary tract infection (Renal and urinary disorders) | 1 (1) — klebsiella pneumoniae urinary tract infection

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-10-28): https://cdn.clinicaltrials.gov/large-docs/79/NCT02936479/Prot_SAP_000.pdf